CLINICAL TRIAL: NCT00272766
Title: Macugen for Histoplasmosis-An Open-Label, Single-Site, Comparative, Prospective Case Series
Brief Title: Macugen for Histoplasmosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Barnes Retina Institute (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0722; 05-1103
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Ocular Histoplasmosis; Choroidal Neovascularization
Keywords: Ocular histoplasmosis; Macugen; Photodynamic therapy with Visudyne; Best-corrected visual acuity scores between 20/40-20/200; classic or occult choroidal neovascularization
MeSH Terms: conditions — Choroidal Neovascularization | interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium

SUMMARY:
The purpose of this study is to evaluate the safety and effect on visual acuity of Macugen (pegaptanib sodium) in patients with subfoveal choroidal neovascularization (CNV) secondary to the ocular histoplasmosis syndrome (OHS).

DETAILED DESCRIPTION:
Ocular histoplasmosis is a leading cause of severe and irreversible central vision loss in middle-aged adults living in the central and eastern US. OHS has been associated with the fungus Histoplasma capsulatum, a dimorphic soil mold found in 18 to 20 states in the central and eastern US. Annually, approximately 100,000 people are thought to be at risk of vision loss caused by OHS.

This study will include OHS patients with CNV lesions no larger than 5400 microns in greatest linear diameter with classic or occult CNV extending under the geometric center of the FAZ and best-corrected visual acuity letter score between 20/40-20/200. Twenty four patients will be enrolled and the study will have 2 treatment arms with 12 patients each. The first arm will consist of 12 patients who will receive 0.3 mg of Macugen intravitreally every 6 weeks for one year. The second arm will consist of 12 patients who will receive Photodynamic Therapy (PDT) with Visudyne every 3 months for one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular histoplasmosis,
* Evidence of classic or occult choroidal neovascularization extending under the geometric center of the fovea,
* Greatest linear diameter of no greater than 5400 microns,
* Best-corrected visual acuity scores between 20/40-20/200,
* Ability to give informed consent,
* Limited child bearing potential and a negative pregnancy test

Exclusion Criteria:

* Features of any condition other than OHS such as AMD, or pathologic or myopic angioid streaks associated with CNV in the study eye,
* Area of CNV that is less than 50% of the total lesion not including area of prior laser treatment, previous rip of retinal pigment epithelium,
* Vitelliform-like lesion,
* Telangiectasia,
* Central serous retinopathy,
* Serous pigment epithelial detachment without CNV,
* Any significant ocular disease other than CNV that could compromise vision in the study eye, such as amblyopia, glaucoma, optic neuropathy, or diabetic retinopathy,
* Inability to obtain photographs to document CNV,
* Presence of atrophy/scar in the center of fovea,
* Presence of vitreo-retinal traction over the center of the fovea,
* History of treatment for CNV in the study eye other than non-foveal laser photocoagulation,within 12 weeks prior to enrollment
* Participation in another clinical trial or use of another investigational new drug within 12 weeks of the full extent of the study treatment,
* Intraocular surgery within the last two months,
* Capsulectomy within the last month in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-02; Study Completion 2007-05

PRIMARY OUTCOMES:
Visual function measurements, including change from baseline in visual acuity: lesion size: and leakage for one year

SECONDARY OUTCOMES:
Patients who gain 7 or more letters or patients who lose 8 or more letters from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav K Shah, MD, Principal Investigator — Barnes Retina Institute
Locations (1):
- Barnes Retina Institute, St Louis, Missouri, United States